CLINICAL TRIAL: NCT06173895
Title: A Phase 1, Open-Label Study to Determine the Relative Bioavailability of LY3454738 in Healthy Participants
Brief Title: A Relative Bioavailability Study of LY3454738 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18391; J1B-MC-FRCJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3454738 (Test Formulation) (Experimental)
  Interventions: Drug: LY3454738
- LY3454738 (Reference Formulation) (Experimental)
  Interventions: Drug: LY3454738

INTERVENTIONS:
Drug: LY3454738 — Administered subcutaneously (SC)

SUMMARY:
The main purpose of this study is to look at the amount of the study drug, LY3454738 that gets into the blood stream and how long it takes the body to get rid of it when given under the skin comparing a test formulation versus a reference formulation in healthy participants. The study will also evaluate the safety and tolerability of LY3454738 and information about any side effects experienced will be collected. For each participant, the total duration of the study will be approximately up to 17 weeks, including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical history and physical examination.
* Have body mass index (BMI) between 18.0 and 28.0 kilograms per meter squared (kg/m²), inclusive, at screening.

Exclusion Criteria:

* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational medicinal product; or of interfering with the interpretation of data.
* Had any surgical procedure (except for minor surgery requiring local or no anesthesia and without any complications or sequelae) within 12 weeks prior to screening or intend to during the study.
* Show evidence of active or latent TB.
* Have one of the following infections: hepatitis B virus or human immunodeficiency virus (HIV).
* Participants must not be currently participating in or completed a clinical trial within the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3454738 | Predose on day 1 up to 85 days post dose
  PK: Cmax of LY3454738
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3454738 | Predose on day 1 up to 85 days post dose
  PK: AUC of LY3454738

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No